CLINICAL TRIAL: NCT01279811
Title: The Canadian Multicentre CSF Monitoring and Biomarker Study
Acronym: CAMPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Rick Hansen Institute (Other)
Responsible Party: Principal Investigator, Brian Kwon, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H10-01091
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury, CSF, biomarkers, CSF pressure
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Vasoconstrictor Agents; Dopamine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): Vasopressor Crossover - Dopamine & NORepinephrine
  Interventions: Other: Crossover of vasopressors

INTERVENTIONS:
Other: Crossover of vasopressors — To evaluate the effect of different vasopressor agents on SCPP, a "crossover" intervention will be conducted on patients requiring either NORepinephrine or DOPamine post-operatively, once daily for 5 days while the catheter is in place. A subject on NORepinephrine will be switched over to DOPamine for 1 hr, and then switched back to NORepinephrine. Likewise, a subject on DOPamine will be switched over to NORepinephrine for 1 hr, and then switched back to DOPamine. Subjects on both vasopressors will have DOPamine stopped for 1 hr and NORepinephrine titrated up to maintain the same MAP for 1 hr, and then brought back to the original levels of both vasopressors. On the following day, the reverse will be carried out, with a stoppage of the NORepinephrine and maintenance solely on DOPamine.
  Other Names: vasopressors; DOPamine; NORepinephrine

SUMMARY:
The purpose of this study is to:

1. Measure the pressure in the spinal fluid surrounding the spinal cord to find out how well the spinal cord is being supplied with blood.
2. Determine how drugs called "vasopressors", which are used to control blood pressure following SCI (spinal cord injury), influence spinal fluid pressure.
3. Characterize the severity of an SCI using the levels of specific proteins found within the spinal fluid.
4. Predict how much neurologic recovery may be regained using the levels of specific proteins within your spinal fluid.
5. Identify proteins within the spinal fluid that will help us learn more about what is happening after SCI and assist us in developing new treatments for SCI.

DETAILED DESCRIPTION:
This research project consists of two complementary yet distinct initiatives:

1. First, we will prospectively evaluate spinal cord perfusion pressure(SCPP)in patients with acute spinal cord injuries, to provide scientifically-based guidelines on the management of blood pressure during the acute injury phase.
2. Second, we will evaluate cerebrospinal fluid(CSF) samples from these patients with the goal of prospectively validating a series of biochemical markers that correlate with injury severity and predict neurologic outcome. Ultimately, our goals are to enhance the neurologic outcome of individuals with spinal cord injuries by improving upon their acute clinical care, and to establish biological surrogates of injury severity that may be used to facilitate clinical trials of novel therapeutic interventions for acute spinal cord injury.

Specific Aims

This multicenter study will enroll patients with acute traumatic cervical and thoracic SCI within 48 hours of their injury. A lumbar intrathecal catheter will be inserted pre-operatively for the measurement of intrathecal pressure (ITP) and the collection of CSF samples. Spinal cord perfusion pressure will be calculated as the difference between mean arterial pressure (MAP) and the ITP. The objectives of this aspect of the study will be to:

* Document the changes in SCPP over the first 5-7 days post-injury (with an intrathecal catheter that is in place for 5 days).
* Determine the effect of different vasopressor agents on SCPP.

Additionally, CSF samples will be obtained from the intrathecal catheter at 8-hour intervals to analyse the expression of the following biochemical markers: including interleukin (IL)-6, IL-8, monocyte chemo-attractant protein (MCP)-1, glial fibrillary acidic protein (GFAP), S100beta, and tau. The objectives of this aspect of the study will be to:

* Evaluate the accuracy of these inflammatory and neuronal markers at classifying the initial severity of paralysis and at predicting the extent of neurologic recovery.
* Characterize the temporal pattern of expression of these proteins to provide a more complete description of the human pathophysiology of SCI.

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age or older
* Complete (AIS A)or incomplete (AIS B, C) acute SCI involving bony spinal levels between C0 and L1
* Non-penetrating injury
* Able to communicate in English and provide informed consent
* Enrolled within 48 hours after injury and able to provide CSF and blood samples within this period

Exclusion Criteria:

* SCI that involves sensory impairment only (i.e., no impairment in ability to move arms and legs)
* Penetrating spinal cord injury
* Isolated radiculopathy (injury only to the nerve outside of the spinal cord)
* Cauda equina injury (injury to nerve roots at the end of the spinal cord)
* Severe injury to head at the time of the SCI
* Injury to lower back (below the spinal level L1)
* Major injury to legs, arms, pelvis, chest, or abdomen that make it impossible for doctors to tell how severely injured the spinal cord is
* Have a pre-existing neurological disorder such as Parkinson's disease, Alzheimer's disease, Huntington's disease, or multiple sclerosis or amyotrophic lateral sclerosis.
* Pre-existing thromboembolic disease or coagulopathy (disorders related to blood clotting), such as haemophilia or von Willebrand's disease
* Pre-existing and ongoing infection in the body (e.g., pneumonia, urinary tract infection, cellulitis)
* Pre-existing inflammatory or autoimmune disorder such as rheumatoid arthritis, systemic lupus, psoriasis
* Systemic disease that may interfere with safety or evaluation of the condition we're studying (e.g., heart disease, HIV, HTLV-1)
* Any other medical condition that in the investigator's opinion would render the study procedures dangerous or impair ability to receive study therapy
* Pregnancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Spinal cord perfusion pressure | 5 days
  SCPP will be calculated as the difference between the MAP and ITP. The ITP and MAP will be recorded over 5 days(5-7 days post-injury) while the lumbar intrathecal catheter is in place.

SECONDARY OUTCOMES:
Levels of specific biochemical markers in the CSF | 5 days
  CSF samples will be obtained from the intrathecal catheter at 8-hour intervals, three times daily for 5 days. These samples will be evaluated will the goal of prospectively validating a series of biochemical markers that correlate with injury severity and predict neurologic outcome.
International Standards for Neurological Classification of Spinal Cord Injury (aka ASIA Examination) | 1 year
  For the purposes of ensuring that neurologic deterioration is not occurring while the lumbar intrathecal catheter is in place, an ASIA assessment will be performed daily while the intrathecal catheter is inserted. For the purpose of documenting neurologic recovery over time, the ASIA examination will also be performed at 3, 6, and 12 months post-injury.
DN4 and other pain questionnaires | 1 year
  It is currently believed that the development of neuropathic pain is closely related to neuroinflammation after SCI. In an effort to determine if we could establish etiologic cytokines, we will administer the DN4 and other pain questionnaires to characterize and quantify neuropathic pain. These questionnaires will be administered at screening, days 1-5 post-insertion of the lumbar intrathecal catheter, 3 months, 6 months and 1 year post-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Brian K. Kwon, MD,PhD, Principal Investigator — University of British Columbia and Vancouver General Hospital
Locations (6):
- Zuckerberg San Francisco General Hospital (UCSF), San Francisco, California, United States
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Health Science Centre- Victoria Campus, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital du Sacré-Coeur, Montreal, Quebec

REFERENCES:
- [Derived] Stukas S, Cooper J, Gill J, Fallah N, Skinnider MA, Belanger L, Ritchie L, Tsang A, Dong K, Streijger F, Street J, Paquette S, Ailon T, Dea N, Charest-Morin R, Fisher CG, Bailey CS, Dhall S, Mac-Thiong JM, Wilson JR, Christie S, Dvorak MF, Wellington CL, Kwon BK. Association of CSF and Serum Neurofilament Light and Glial Fibrillary Acidic Protein, Injury Severity, and Outcome in Spinal Cord Injury. Neurology. 2023 Mar 21;100(12):e1221-e1233. doi: 10.1212/WNL.0000000000206744. Epub 2023 Jan 4. PMID 36599698
- [Derived] Rosner J, Negraeff M, Belanger LM, Tsang A, Ritchie L, Mac-Thiong JM, Christie S, Wilson JR, Dhall S, Charest-Morin R, Street J, Ailon T, Paquette S, Dea N, Fisher CG, Dvorak MF, Finnerup NB, Kwon BK, Kramer JLK. Characterization of Hyperacute Neuropathic Pain after Spinal Cord Injury: A Prospective Study. J Pain. 2022 Jan;23(1):89-97. doi: 10.1016/j.jpain.2021.06.013. Epub 2021 Jul 21. PMID 34302956